CLINICAL TRIAL: NCT01374919
Title: Total Dose Infusion of Ferumoxytol (1020mg) in 15 Minutes for Iron Defeciency Anemia
Brief Title: Total Dose Infusion of Ferumoxytol(1020mg) in 15 Minutes for Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auerbach Hematology Oncology Associates P C (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Auerbach MD, Principal Investigator, Auerbach Hematology Oncology Associates P C
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ferumoxytol 1020
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Iron Deficiency Anemia
Keywords: Intravenous iron; ferumoxytol; iron deficiency anemia; Treatment of iron deficiency; Intolerance of or ineffectiveness of oral iron
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ferumoxytol (Other): IV administration of 1020 mg of ferumoxytol in 15 minutes
  Interventions: Drug: ferumoxytol

INTERVENTIONS:
Drug: ferumoxytol — IV administration of 1020 mg of ferumoxytol in 15 minutes
  Other Names: Feraheme, intravenous iron, total dose infusion

SUMMARY:
The aim of the study is to recruit 30 patients who have been referred to Auerach Hematology Oncology Assoc. for the treatment of iron defeciency anemia with iv iron (Ferumoxytol 1020 mg) administered via infusion pump over 15 minutes.

To ascertain acute safety and tolerability of ferumoxytol during immediate post dosing observation period.

Assess additional safety profile and laboratory assessment at follow up visit and interim telephone follow up.

DETAILED DESCRIPTION:
Ferumoxytol, a modified iron dextran, which allows the rapid administration of IV iron without free iron release, was approved for a 510 mg injection to be administered in not less than 17 seconds. Although this represents a felicitous treatment for patients who come frequently, such as dialysis and chemotherapy patients, multiple publications suggest that full dose replacement is usually at the 1000 mg level. No studies extant are available with this dosing schedule for ferumoxytol. In this trial, iron deficient patients with hemoglobin levels of <11.0 grams per deciliter will be consented to received 1020 mg (two 510 mg vials) of ferumoxytol in 15 minutes. Vital signs will be performed at 5, 10, 15, 30 and 60 minutes. Followup phone calls for any clinical adverse events will be made at 24-48 hours and one week after administration. At four weeks follow-up hematologic and serologic (iron parameters) will be made along with a physician visit.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficiency anemia intolerant of or failure to respond to oral iron or condition where oral iron is known to be ineffective or harmful.
* Subject must be able to be contacted at 24-48 hours after dose and come for followup at four weeks.
* Subject must be capable of understanding informed consent
* No other form of iron may be taken within four weeks of consent or for four weeks after treatment

Exclusion Criteria:

* History of hypersensitivity to ferumoxytol.
* Imminent dialysis.
* Anemia due to other etiology.
* Parenteral iron within 4 weeks of consent.
* Pregnancy.
* Erythropoiesis stimulating agent within 30 days of consent.
* Other illness that would interfere with participation or understanding of trial.
* Major surgery planned within four weeks of consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Auerbach, MD, Principal Investigator — Auerbach Hematology and Oncology
Locations (1):
- Auerbach Hematology and Oncology, Baltimore, Maryland, United States

REFERENCES:
- [Result] Auerbach M, Strauss W, Auerbach S, Rineer S, Bahrain H. Safety and efficacy of total dose infusion of 1,020 mg of ferumoxytol administered over 15 min. Am J Hematol. 2013 Nov;88(11):944-7. doi: 10.1002/ajh.23534. Epub 2013 Sep 9. PMID 23828252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from routine referrals from obgyns, gastroenterologists, bariatric surgeons, general internists and nephrologists. All patients were iron deficient and anemic. All were oral iron intolerant. The data were presented at the 2012 American Society of Hematology meeting.
Groups:
- Total Dose 1020 mg Feramoxytol: All participants receive 1020 mg of Feramoxytol.
Period: Overall Study
Arm/Group | Total Dose 1020 mg Feramoxytol
Started | 60
Completed | 58
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Dose 1020 mg Feramoxytol
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 53.4 (67) [22 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of 1020 mg of Ferumoxytol Over 15 Minutes. Hemoglobin Measurements Will Take Place at Four and Eight Week Visit.
Description: Percentage of participates with indicated increase in hemoglobin from baseline to week 4 and week 8
Time Frame: baseline 4 weeks and 8 weeks
Population: Two patients had minor infusion reactions and refused rechallenge. All other patients completed the study. Their hemoglobin levels, the primary outcome, were obtained at 4 and 8 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Total Dose 1020 mg Feramoxytol
Number analyzed (Participants) | 58
percentage of participants
  Greater than 1 g/dl increase at week 4 | 85
  Greater than 2 g/dl at week 4 | 58
  Greater than 1 g/dl increase at week 8 | 92
  Greater than 2 g/dl increase at week 8 | 86

2. Secondary Outcome: Number of Participants With Treatment Related Serious Adverse Events. Calls for Minor Side Effects Will Occur at 24 and 48 Hours and One Week. A Followup Visit Will Occur at 4 Weeks.
Time Frame: immediate, 24 and 48 hours, one week and followup visit at 4 weeks
Measure: Number; unit: participants
Arm/Group | Total Dose 1020 mg Feramoxytol
Number analyzed (Participants) | 60
participants | 0

ADVERSE EVENTS:
Time Frame: 8 weeks from treatment day
Description: Patients were observed for one hour after administration. Telephone calls were made at 24 and 48 hours and 7 days for delayed AEs. Follow visits in the office occurred at 4 and 8 weeks.
Arm/Group | Total Dose 1020 mg Feramoxytol
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 22/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Dose 1020 mg Feramoxytol (N=60)
Arthralgia/Myalgia/Muscle Spasm (Musculoskeletal and connective tissue disorders) | 14
Headache (Musculoskeletal and connective tissue disorders) | 8
Chest Pressure (Musculoskeletal and connective tissue disorders) | 4
Pruritis (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 — Unrelated to drug
Flushing (General disorders) | 3
abdominal pain (Gastrointestinal disorders) | 2 — Unrelated to drug
Fever (General disorders) | 1
dry mouth (Gastrointestinal disorders) | 1 — unrelated to drug
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
edema (General disorders) | 1
metallic taste (General disorders) | 1
lip swelling (Immune system disorders) | 1
nausea (Gastrointestinal disorders) | 3
dizziness (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No